CLINICAL TRIAL: NCT01227382
Title: Prospective Evaluation of the Accuracy of Spybite Biopsy Forceps for the Tissue Diagnosis of Lesion of the Pancreatobiliary System. ( Part of the "The Clinical Utility of Cholangioscopy and Pancreatoscopy in the Diagnosis and Treatment of Pancreaticobiliary Disorders" Study)
Brief Title: Accuracy of Spybite Forceps When Compared to Conventional Sampling Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SpyBite
Record Dates: First submitted 2010-10-18; First posted 2010-10-25 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Accuracy of Tissue Diagnosis; Bile Duct Stricture; Pancreatic Duct Stricture
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ERCP with Cholangiopancreatoscopy (Other): The subjects who have been scheduled for an Endoscopic Retrograde Cholangiopancreatography (ERCP) with Cholangiopancreatoscopy for evaluation of a bile duct or pancreatic duct stricture sampling.
  Interventions: Procedure: ERCP with cholangiopancreatoscopy

INTERVENTIONS:
Procedure: ERCP with cholangiopancreatoscopy — Endoscopic Retrograde Cholangiopancreatography (ERCP)with cholangiopancreatoscopy and sampling of stricture with SpyBite biopsy forceps, cytology brush and RJ3biopsy forceps
  Other Names: Endoscopic Retrograde Cholangiopancreatography; ERCP

SUMMARY:
The investigators are evaluating the use of a SpyBite biopsy forceps for tissue diagnosis when compared to standard biopsy techniques.

DETAILED DESCRIPTION:
The participants will undergo an Endoscopic Retrograde Cholangiopancreatography (ERCP) with cholangiopancreatoscopy and evaluation of a bile duct or pancreatic duct stricture with three different types of techniques for biopsy: SpyBite biopsy forceps, cytology brush and RJ3biopsy forceps.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects is 18 years or older
2. Scheduled to undergo Endoscopic Retrograde Cholangiopancreatography (ERCP) wiht cholangioscopy and/or pancreatoscopy at the University of Florida Gainesville Florida as medically indicated.
3. Lesion of the pancreatobiliary system that requires tissue sampling as medically indicated
4. Subject myst be able to give informed consent

Exclusion Criteria:

1. Any contraindication to Endoscopic Retrograde Cholangiopancreatography (ERCP)
2. The subject is unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Flordia
Locations (1):
- Shands at UF Ensopcopy, Gainesville, Florida, United States

REFERENCES:
- [Derived] Draganov PV, Chauhan S, Wagh MS, Gupte AR, Lin T, Hou W, Forsmark CE. Diagnostic accuracy of conventional and cholangioscopy-guided sampling of indeterminate biliary lesions at the time of ERCP: a prospective, long-term follow-up study. Gastrointest Endosc. 2012 Feb;75(2):347-53. doi: 10.1016/j.gie.2011.09.020. PMID 22248602

RESULTS

PARTICIPANT FLOW:
Groups:
- Indeterminate Biliary Lesions Requiring Tissue Sampling: Each patient underwent triple sampling of the identified biliary lesion with cholangioscopy-guided mini-forceps biopsy, standard cytology brushing, and standard forceps biopsy.
Period: Overall Study
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.92 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Accurate Diagnoses of Cancer
Description: The diagnostic accuracy of the Spybite Biopsy forceps was compared to both the cytology brush and the RJ3 biopsy forceps sampling of any stricture or biliary lesions found on Endoscopic Retrograde Cholangiopancreatography (ERCP). All three methods were used at baseline to obtain a sample for the determination of cancer vs. no cancer.
Time Frame: up to 7 days after the procedure
Population: Percentage of participants with accurate diagnoses of cancer
Measure: Number; unit: percentage of accurate diagnoses
Groups:
- Diagnostic Accuracy of SpyBite Biopsy Forceps Compared to the: Each patient underwent triple sampling of the identified biliary lesion or stricture with cholangioscopy-guided Spybite forceps biopsy, standard cytology brushing, and standard forceps biopsy.
Arm/Group | Diagnostic Accuracy of SpyBite Biopsy Forceps Compared to the
Number analyzed (Participants) | 26
percentage of accurate diagnoses
  Cytology brush | 38.5
  Standard forceps biopsy | 53.9
  Spybite biopsy | 84.6

2. Secondary Outcome: Procedure Technical Success
Description: The procedure technical success was defined when all of the following criteria were met: Successful advancement of the cholangioscope to the desired target, adequate cholangioscopic visualization of the area of interest, and successful applications of of all sampling maneuvers with visible tissue seen macroscopically when obtaining mini forceps and standard forceps biopsy samples.
Time Frame: day 1
Population: Percentage of participants with accurate diagnoses of cancer
Measure: Number; unit: participants
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Number analyzed (Participants) | 26
participants | 26

3. Secondary Outcome: Total Procedure Time
Description: The total time to perform ERCP
Time Frame: 120 minutes
Population: Percentage of participants with accurate diagnoses of cancer
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Indeterminate Biliary Lesions Requiring Tissue Sampling: Each patient underwent triple sampling of the identified biliary lesion or stricture with cholangioscopy-guided Spybite forceps biopsy, standard cytology brushing, and standard forceps biopsy.
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Number analyzed (Participants) | 26
minutes | 54.00 (12.71)

4. Secondary Outcome: Total Cholangioscopy Time
Description: This is the total time it takes for the dye to be performed during the ERCP.
Time Frame: 60 minutes
Population: Percentage of participants with accurate diagnoses of cancer
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Number analyzed (Participants) | 26
minutes | 23.65 (9.43)

5. Secondary Outcome: Cholangioscopy Visualization Time
Description: The portion of the total ERCP time spent on Cholangioscopy visualization.
Time Frame: 30 minutes
Population: Percentage of participants with accurate diagnoses of cancer
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Number analyzed (Participants) | 26
minutes | 11.69 (8.03)

6. Secondary Outcome: Sampling Times for Each Device
Description: The sampling time of the Spybite Biopsy forceps was compared to both the cytology brush and the RJ3 biopsy forceps of any stricture or biliary lesions found on Endoscopic Retrograde Cholangiopancreatography (ERCP).
Time Frame: 15 minutes
Population: Percentage of participants with accurate diagnoses of cancer
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Number analyzed (Participants) | 26
minutes
  Spybite forceps | 11.92 (4.67)
  Standard cytology brushing | 3.77 (1.21)
  Standard forceps biopsy | 5.73 (3.11)

7. Secondary Outcome: Adverse Events
Description: Adverse events were prospectively evaluated at the end of the procedure, at discharge from the endoscopy unit, and by telephone call 24 hours post procedure. Adverse events were defined and graded using the 2010 American Society for Gastrointestinal Endoscopy consensus criteria.
Time Frame: 24 hours
Population: Percentage of participants with accurate diagnoses of cancer
Measure: Number; unit: participants
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Number analyzed (Participants) | 26
participants | 3

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Indeterminate Biliary Lesions Requiring Tissue Sampling
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 2/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indeterminate Biliary Lesions Requiring Tissue Sampling (N=26)
Postsphincterotomy Bleeding (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indeterminate Biliary Lesions Requiring Tissue Sampling (N=26)
Mild Pancreatitis (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes